CLINICAL TRIAL: NCT05511831
Title: A Randomized Controlled Study on the Efficacy and Safety of Ketotifen in Primary PCI Patients With STEMI
Brief Title: The Efficacy and Safety of Ketotifen in Primary PCI Patients With STEMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2022319
Record Dates: First submitted 2022-08-19; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
Keywords: ketotifen; STEMI; mast cell; prognosis
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Ketotifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketotifen (Experimental): Ketotifen was added to the standard treatment within 24 hours after the completion of primary PCI for 3 months, taking 1 mg each time, 1-2 times a day according to the patient's tolerance.
  Interventions: Drug: Ketotifen Fumarate
- Control group (Sham Comparator): Standard treatment according to guidelines
  Interventions: Drug: standard treatment

INTERVENTIONS:
Drug: Ketotifen Fumarate — Ketotifen treatment for 3 months, 1 mg each time, 1-2 times a day according to the patient's tolerance
  Other Names: Ketotifen
  Arms: ketotifen
Drug: standard treatment — Standard treatment methods will be determined according to the Guidelines for the Diagnosis and Treatment of Acute ST-segment Elevation Myocardial Infarction (2019) [19], including primary PCI, dual antiplatelet, anticoagulation, ACEI/ARB/ARNI, β-receptor blockade drugs, statins, etc.
  Other Names: standard
  Arms: Control group

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of ketotifen (MC stabilizer) on the basis of standard treatment after primary PCI in STEMI patients. The ketotifen group and the control group were the ketotifen group and the control group. The control group continued to receive STEMI standard treatment. The ketotifen group received ketotifen for 3 months on the basis of standard treatment within 24 hours after primary PCI, and was followed up for 1 year. Infarct size, as well as differences in echocardiography, markers of two-dimensional speckle tracking, inflammatory factors and MC markers, and major adverse cardiovascular events.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) is the best way to improve the prognosis of patients with acute ST-segment elevation myocardial infarction (STEMI). However, STEMI after PCI may still have ischemia-reperfusion injury, inappropriate ventricular remodeling and myocardial fibrosis, which may be related to the inflammatory response of STEMI. Mast cells (MCs) and their degranulation products play an important role in the inflammatory response as well as inducing a series of inflammatory factors. It has been observed in animal experiments that MC stabilizers can improve the ejection fraction, reduce myocardial infarction size and myocardial fibrosis in patients with STEMI, but there is a lack of clinical studies to confirm the role of MC stabilizers in STEMI. The purpose of this study was to evaluate the efficacy and safety of ketotifen (MC stabilizer) on the basis of standard treatment after primary PCI in STEMI patients. The ketotifen group and the control group were the ketotifen group and the control group. The control group continued to receive STEMI standard treatment. The ketotifen group received ketotifen for 3 months on the basis of standard treatment within 24 hours after primary PCI, and was followed up for 1 year. Infarct size, as well as differences in echocardiography, markers of two-dimensional speckle tracking, inflammatory factors and MC markers, and major adverse cardiovascular events, to demonstrate that ketotifen can reduce ischemia-reperfusion injury and improve ventricular reperfusion in AMI. It provides new ideas for the treatment of AMI and a new basis for the optimization of STEMI treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Ages above 18 and below 80, gender is not limited;
* Meet the diagnostic criteria for STEMI (diagnostic criteria: ischemic chest pain lasting ≥30 min; ST segment elevation in two or more adjacent leads on the ECG or new left bundle branch block; with or without elevation of myocardial markers) , have completed primary PCI, and received standard treatment according to the Chinese "Guidelines for the Diagnosis and Treatment of Acute ST-segment Elevation Myocardial Infarction (2019)", including dual antiplatelet, anticoagulation, beta receptor Blockers, statins, etc.
* No contraindications to ketotifen;
* Agree and cooperate with participating in this research.

Exclusion Criteria:

* Severe heart failure, such as Killip grade III-IV or LVEF <35%;
* Coronary artery bypass grafting within the past 3 years or planned;
* The patient is using or planning to use long-term oral or intravenous glucocorticoids (inhaled and topical hormones are allowed);
* Patients with severe liver and kidney disease;
* Patients with a history of cancer or lymphoproliferative diseases in the past 3 years;
* Implanted metal in the body or claustrophobia cannot accept cardiac MRI;
* Pregnancy or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Myocardial infarct size | 3 months after myocardial infarction
  Myocardial infarct size was assessed by cardiac MRI

SECONDARY OUTCOMES:
left ventricular systolic function | 24 hours, 1 month, 3 months, and 12 months after myocardial infarction
  Transthoracic echocardiography to measure LVEF, left ventricular end-diastolic diameter, Em/Sm
Left ventricular ultrasound strain | 24 hours, 1 month, 3 months, and 12 months after myocardial infarction
  Two-dimensional speckle tracking imaging measures the movement in the long-axis direction as the overall longitudinal strain, the movement in the short-axis direction as the overall radial strain, reflecting the degree of wall systolic thickening, and the annular motion in the short-axis direction as the overall circumferential strain
inflammatory factors and MC markers | 24 hours, 1 month, 3 months, and 12 months after myocardial infarction
  Analysis of inflammatory factors (such as TNF-α, IL1, IL6, etc.) and MC markers (chymotrypsin)
major adverse cardiovascular events | 12 months
  MACE events (death, nonfatal myocardial infarction, unplanned revascularization, hospitalization for angina and readmission for heart failure)
Drug-Related Adverse Reactions | 12 months
  Fatigue, lethargy and lethargy, nausea and other gastrointestinal adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Ming Cui, Doctor, Study Director — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No